CLINICAL TRIAL: NCT01908920
Title: Osteopathic Manipulative Treatment Effects on High Frequency Parameters in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute for Evidence Based Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Francesco Cerritelli, MS, DO, European Institute for Evidence Based Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HRVOST
Record Dates: First submitted 2013-07-19; First posted 2013-07-26 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Healthy Subject; Heart Rate Variability
MeSH Terms: interventions — Manipulation, Osteopathic; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OMT (Other): Each osteopathic session is based on structural evaluation and treatment using indirect techniques.
  Interventions: Other: Osteopathic manipulative treatment
- SHAM (Other): Sham therapy was administered with subjects lying supine on the treatment table while the operator used light manual contact to "treat" the subject. A pre-determined protocol has been used. The practitioner's attention was distracted by subtracting calculation in silence.
  Interventions: Other: SHAM
- CONTROL (Other): No intervention
  Interventions: Other: CONTROL

INTERVENTIONS:
Other: Osteopathic manipulative treatment
  Arms: OMT
Other: SHAM
  Arms: SHAM
Other: CONTROL
  Arms: CONTROL

SUMMARY:
The aim of the present study is to determine the extend to which osteopathic manipulative treatment (OMT) is effective on a sample of healthy subjects in changing high frequency (HF) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45;
* No chronic symptomatology;
* No acute symptomatology during the last 72 hours before intervention;
* No pathologies

Exclusion Criteria:

* Age below 18 or over 45;
* Pregnancy;
* Menopause;
* Abuse of alcool during the last 48 hours;
* Chronic pain;
* Acute pain during the last 72 hours;
* Conclamate pathologies;
* Use of drugs during the last 72 hours ;
* Use of ortothic devices during the last 3 months;
* Any type of surgery;
* Osteopathic treatment during the last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline high frequency (HF) value at 1 week | baseline and 1 week

SECONDARY OUTCOMES:
Change from baseline in low frequency (LF) value at 1 week | baseline and 1 week
Change from baseline LF/HF ratio value at 1 week | baseline and 1 week
Change from baseline very low frequency (VLF) value at 1 week | baseline and 1 week
Change from baseline standard deviation beat-to-beat (SDNN) value at 1 week | baseline and 1 week
Changes from baseline square root of the mean squared difference of successive beat-to-beat (RMSSD) at 1 week | baseline and 1 week
Change from baseline proportion of beat-to-beat50 divided by total number of beat-to-beats in (pNN50) at 1 week | baseline and 1 week
Change from baseline detrended fluctuation scaling exponent (DFAa1) value at 1 week | baseline and 1 week
Change in LF value | during treatment session
Change in LF/HF ratio value | during treatment session
Change in VLF value | during treatment session
Change in SDNN value | during treatment session
Change in RMSSD value | during treatment session
Change in pNN50 value | during treatment session
Change in DFAa1 value | during treatment session
Change from baseline intrasubject HF value at 1 week | baseline and 1 week
Change from baseline heart rate variability parameters between smokers and no-smokers at 1 week | baseline and 1 week
Change from baseline 15D questionnaire at 1 week | baseline and 1 week
Differences in skin conductance value between groups | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, MS, DO, Study Chair — Italian Academy of Traditional Osteopathy - AIOT
Locations (1):
- Accademia Italiana Osteopatia Tradizionale, Pescara, Italy

REFERENCES:
- [Derived] Ruffini N, D'Alessandro G, Mariani N, Pollastrelli A, Cardinali L, Cerritelli F. Variations of high frequency parameter of heart rate variability following osteopathic manipulative treatment in healthy subjects compared to control group and sham therapy: randomized controlled trial. Front Neurosci. 2015 Aug 4;9:272. doi: 10.3389/fnins.2015.00272. eCollection 2015. PMID 26300719